CLINICAL TRIAL: NCT02694445
Title: Monetary Cost of Alzheimer's Disease in China: Study Protocol for a Cluster Randomized Observational Study
Brief Title: Monetary Cost of Alzheimer's Disease in China
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Chinese Medical Doctor Association (Other)
Responsible Party: Principal Investigator, Jianping Jia, Professor, Beijing Friendship Hospital
Other Study IDs: MAC-001
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: observation — The study is non-interventional.

SUMMARY:
The purpose of the study is to estimate the Chinese economic burden in patients with Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This observational study covered all the 30 provincials/municipals/autonomous in mainland China except Hong Kong and Macau. Tier 3 hospitals, psychiatric hospitals, elderly hospitals, nursing home and communities were randomly selected as research centers, and more than 2500 patients with AD and their caregivers were enrolled at last. The main outcome of this study was assessed not only by the electronic medical system of communities and hospitals, but also by questionnaires. Using a societal prevalence-based gross COI approach to estimated the total yearly costs of AD in China.

ELIGIBILITY:
Inclusion Criteria:

1. New patients who are diagnosed with AD in this investigation or old patients who were diagnosed prior to this investigation were eligible；
2. AD diagnosis must meet criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and the National Institute of Neurologic and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA). The diagnosis should also meet the following: Modified Hachinski Ischemic Scale (MHIS) score≤4, Activity of Daily Living Scale (ADL) score≥23, Geriatric Depression Scale (GDS) score<11. Neuroimaging MRI support AD diagnosis (exist atrophy in medial temporal lobe, white matter lesions score≤2 minutes according to the Fazekas criteria. AD disease classification according to mini-mental state examination (MMSE) scale (for illiterate dementia: mild: 21~24 points; moderate: 11~20 points; severe: 10 points or less; for lettered dementia: mild: 16~19 points; moderate: 8~15 points; severe: 7 points or less). The diagnosis of AD was confirmed by brain CT or MRI scans and by laboratory tests to rule out any other significant comorbidity.
3. 60-year-old and above, men or women.
4. Normal vision or corrected visual, normal audition or corrected auditory, and cooperate with inspections and treatments.
5. Consent to participate with a signed informed consent by himself/herself or guardians.

Exclusion Criteria:

1. Patient with vascular dementia or dementia caused by other reasons, such as major depression or other major psychiatric illnesses, thyroid dysfunction, encephalitis, multiple sclerosis, and other dementia which includes frontotemporal dementia (FTD), dementia with Lewy bodies (DLB), and Parkinson's dementia (PDD).
2. MRI and laboratory tests (blood cell counts, liver and renal function, electrolyte, vitamin B12/folic, HIV, syphilis, and so on) do not support or rule out AD diagnoses.
3. Has a history of alcoholism and drug abuse.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzhemer's disease and their caregivers.
Sampling Method: Probability Sample
Enrollment: 3098 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Jianping, Doctor, Study Chair — Head of Neurology Department, Capital Medical University
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li F, Chen S, Wei C, Jia J. Monetary costs of Alzheimer's disease in China: protocol for a cluster-randomised observational study. BMC Neurol. 2017 Jan 25;17(1):15. doi: 10.1186/s12883-017-0802-9. PMID 28122529

RESULTS

PARTICIPANT FLOW:
Groups:
- Participant Patients: Patient aged ≥60 years, inclusion criteria were: (1) a primary diagnosis of AD according to the National Institute of Neurologic and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria, 13 diagnosed by a dementia specialist; (2) complete information about the economic costs of AD and comorbidities, obtained from electronic medical records systems and face-to-face interviews; and (3) no co-morbidity with direct medical cost > 10% of the total annual costs due to AD.
Period: Overall Study
Arm/Group | Participant Patients
Started | 3098
Completed | 3046
Not Completed | 52

BASELINE CHARACTERISTICS:
Arm/Group | Participant Patients
Number analyzed (Participants) | 3046
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.24 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1651
  Male | 1395
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 3046

OUTCOME MEASURES:

1. Primary Outcome: The Annual National Total Socioeconomic Cost for All AD Patients in China
Description: The annual national total socioeconomic cost for all patients with AD in China in 2015 was obtained, with the average annual cost per patient with AD from our results multiplied by the all number of patients with AD in 2015. So, the value reported in the data table below represents the total cost for all all participants in China.
Time Frame: one year
Measure: Number; unit: billion US$
Groups:
- Participant AD Patients: Patient aged ≥60 years, inclusion criteria were: (1) a primary diagnosis of AD according to the National Institute of Neurologic and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria, 13 diagnosed by a dementia specialist; (2) complete information about the economic costs of AD and comorbidities, obtained from electronic medical records systems and face-to-face interviews; and (3) no co-morbidity with direct medical cost > 10% of the total annual costs due to AD.
Arm/Group | Participant AD Patients
Number analyzed (Participants) | 3046
billion US$ | 167.74

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious, and other (not including serious) adverse events were not monitored/assessed.
Description: All-cause mortality, serious, and other (not including serious) adverse events were not monitored/assessed.
Arm/Group | Participant Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes